CLINICAL TRIAL: NCT02570490
Title: A Randomized, Double-blind, Multi-center Study to Evaluate the Safety and Efficacy of Oral Sodium Fusidate (CEM-102) Compared to Oral Linezolid in the Treatment of Acute Bacterial Skin and Skin Structure Infections
Brief Title: Oral Sodium Fusidate (CEM-102) Versus Oral Linezolid for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arrevus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE06-301
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2017-06

CONDITIONS: Acute Bacterial Skin and Skin Structure Infections
Keywords: fusidic acid; skin infection
MeSH Terms: conditions — Cellulitis | interventions — Fusidic Acid; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CEM-102 (Sodium fusidate) (Experimental): 1500 mg by mouth every 12 hours for 2 doses, then 600 mg by mouth every 12 hours thereafter, until end of therapy (10 days total)
  Interventions: Drug: sodium fusidate
- Linezolid (Active Comparator): 600 mg by mouth every 12 hours for 10 days
  Interventions: Drug: linezolid

INTERVENTIONS:
Drug: sodium fusidate
  Other Names: CEM-102
  Arms: CEM-102 (Sodium fusidate)
Drug: linezolid
  Arms: Linezolid

SUMMARY:
Phase 3, randomized, double-blind, multi-center efficacy and safety study to evaluate an oral CEM-102 loading dose regimen compared to oral linezolid in the treatment of subjects with ABSSSI

DETAILED DESCRIPTION:
The primary objective is to demonstrate the non-inferiority of oral CEM-102 (loading dose regimen of 1500 mg every 12 hours for 2 doses, followed by 600 mg every 12 hours thereafter) compared to oral linezolid (600 mg every 12 hours), each administered for 10 days, for Early Clinical Response (ECR) in the intent to treat (ITT) analysis set in subjects with acute bacterial skin and skin structure infections (ABSSSI). Subjects with an ABSSSI caused by suspected or documented Gram-positive pathogen(s) at baseline will be randomized 1:1 to study treatment

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 12 to 18 years old must weigh >60 kg
* Patients diagnosed with ABSSSI with at least one systemic sign of infection
* Diagnosed with cellulitis, major cutaneous abscess, or wound infections (traumatic or surgical)
* Surface redness, edema or induration must be of a minimum surface area of 75 cm2, or extending ≥5 cm from the peripheral margin of the abscess
* Suspected or documented ABSSSI caused by a Gram-positive pathogen

Exclusion Criteria:

* Involving a chronic diabetic foot infection (diabetic foot ulcer)
* Involving burns
* Involving an anatomical location (e.g. perirectal area) where the incidence of Gram-negative and/or anaerobic pathogen involvement is likely
* Documented bacteremia associated with the current ABSSSI
* Known severe renal impairment, as indicated by estimated CrCl <30 mL/min (by Cockcroft-Gault calculation)
* Evidence of significant liver disease: ALT >3x ULN, or direct bilirubin >ULN; known cirrhosis with decompensation (i.e. Child-Pugh Class B or C disease)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a response for Early Clinical Response | 48 to 72 hours after starting treatment
  Proportion of subjects with a response for Early Clinical Response (ECR), defined as alive and achieved ≥ 20% reduction from baseline in the lesion size at 48-72 hours after start of study drug, without receipt of additional non-study antibiotic therapy.

SECONDARY OUTCOMES:
Proportion of subjects with clinical success at Post-treatment Evaluation | 7 to 14 days after end of treatment
  Proportion of subjects with clinical success at PTE, in the ITT and clinically evaluable (CE) analysis sets.
Incidence of adverse events [Safety and tolerability], Clinical Laboratory Evaluations | Up to 24 months
  Incidence of adverse events, vital sign changes, physical exam changes, and clinical laboratory evaluations will be presented by study arm

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pushkin, MD, Study Director — Melinta Therapeutics, Inc.
Locations (50):
- United States (49):
  - Anaheim, California
  - Bakersfield, California
  - Buena Park, California
  - Fountain Valley, California
  - La Mesa, California
  - La Palma, California
  - Long Beach, California
  - Los Angeles, California
  - Modesto, California
  - National City, California
  - Oceanside, California
  - Riverside, California
  - San Diego, California
  - San Dimas, California
  - Stockton, California
  - Sylmar, California
  - DeBary, Florida
  - DeLand, Florida
  - Doral, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Orlando, Florida
  - South Miami, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Baker, Louisiana
  - Eunice, Louisiana
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Royal Oak, Michigan
  - St Louis, Missouri
  - Butte, Montana
  - Lincoln, Nebraska
  - Somers Point, New Jersey
  - Teaneck, New Jersey
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Lancaster, South Carolina
  - Summerville, South Carolina
  - Rapid City, South Dakota
  - Jackson, Tennessee
  - Gonzales, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Splendora, Texas
- San Juan, Puerto Rico